CLINICAL TRIAL: NCT05985681
Title: A Dose Escalation Phase I Trial of the Safety and Immunogenicity of RG1-VLP, A Candidate Broadly Protective Vaccine for the Prevention of HPV-Associated Cancer
Brief Title: Testing RG1-VLP Vaccine to Prevent HPV-related Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2023-05780; NCI-2023-05780 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01CN45009-45; UWI20-04-01 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); UWI20-04-01 (Other: DCP); P30CA014520 (NIH); UG1CA242635 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (RG1-VLP, Gardasil-9) (Experimental): Patients receive RG1-VLP IM for 3 doses at months 0, 2, and 6 in the absence of unacceptable toxicity. Patients may also receive Gardasil-9 via injection for 3 doses at 6 months after the 3rd study vaccination (month 12), then at months 14 and 18 in the absence of unacceptable toxicity. Patients also undergo blood sample collection on study and may undergo vaginal swab collection on study.
  Interventions: Procedure: Biospecimen Collection; Biological: HPV16 RG1 VLP Vaccine; Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample and vaginal swab collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: HPV16 RG1 VLP Vaccine — Given IM
  Other Names: 16L1-16L2aa17-36-based Vaccine; HPV16 RG1-VLP; HPV16-RG1VLPs; RG1-VLP Vaccine; RG1-VLPs
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given via injection
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of RG1-virus-like particle (VLP) in preventing human papillomavirus (HPV)-related cancers in women. RG1-VLP is a vaccine that aims to protect against rare HPV types not targeted by currently approved HPV vaccines. HPV is a common sexually-transmitted infection that can cause certain genital and oral cancers. RG1-VLP contains a protein of HPV type 16 (HPV16) with a slightly different structure than the licensed Gardasil-9 vaccine. Gardasil-9 is approved by the Federal Drug Administration to help protect against diseases caused by some types of HPV. Gardasil-9 also contains 9 different HPV proteins. Both vaccines contain alum to stimulate the immune system. The usual approach for the prevention of HPV-related cancers for patients who are at increased risk is to consider the currently approved HPV vaccine like Gardasil-9, as well as to be followed closely by their doctor to watch for the development of cancer via routine pap smears. This trial may allow researchers to find out whether the RG1-VLP vaccine can safely trigger an immune response against HPV in healthy women and if it is better or worse than the usual approach for the prevention of HPV-related cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety of RG1-virus-like particles (VLP) in healthy 18-60 years old women at 3 escalating doses.

SECONDARY OBJECTIVES:

I. Determine the immunogenicity of RG1-VLP in healthy 18-60 year old women at 3 escalating doses via the following assays:

Ia. Determine serum antibody responses induced by RG1-VLP vaccination by both human papillomavirus (HPV) 16 L1 VLP and HPV16 L2 RG1-peptide enzyme-linked immunosorbent assay (ELISA). This will be assessed at months 0, 1, 2, 3, 6, 7 and 12; Ib. Determine whether vaccination-induced serum antibody response neutralizes HPV16. This will be assessed at months 0, 1, 2, 3, 6, 7 and 12.

EXPLORATORY OBJECTIVES:

I. Determine whether vaccination-induced serum antibody response broadly neutralizes high risk (hr) HPV other than HPV16. This will be assessed at months 0, 1, 2, 3, 6, 7 and 12.

II. Determine whether vaccination induces a cell-mediated immune (CMI) response. Peripheral blood mononuclear cells (PBMC) will be isolated at months 0, 1 and 7.

III. Determine whether vaccination-induced serum antibody response upon passive transfer to naive animals, protects mice against hrHPV pseudovirion (PsV) challenge. This will be assessed at months 0 and 7.

IV. Determine whether vaccination results in changes in local antibody titers in vaginal and oral secretions (via oral rinse) and the effects of vaccination on HPV types in optionally-collected vaginal and oral secretions and eyebrow hair samples between months 0, 7 and 12.

V. Assess the safety of recombinant human papillomavirus nonavalent vaccine (Gardasil-9) in healthy women post-administration of RG1-VLP.

OUTLINE: This is a dose-escalation study of RG1-VLP.

Patients receive RG1-VLP intramuscularly (IM) for 3 doses at months 0, 2, and 6 in the absence of unacceptable toxicity. Patients may also receive Gardasil-9 via injection for 3 doses at 6 months after the 3rd study vaccination (month 12), then at months 14 and 18 in the absence of unacceptable toxicity. Patients also undergo blood sample collection on study and may undergo vaginal swab collection on study.

After completion of study treatment, patients are followed up to 6 months post-3rd RG1-VLP vaccination injection or up to 14 days post-3rd Gardasil-9 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 18 - 60 years. Because no dosing or adverse event (AE) data is currently available for the use of RG1-VLP in humans, children and adolescents are excluded from this study
* White blood cell (WBC) between 3000/mm^3 - institutional upper limit of normal
* Hemoglobin (Hgb) between 10 g/dl - institutional upper limit of normal
* Platelets >= 100,000/mm^3
* Serum creatinine within institutional normal limits
* Bilirubin =< 2x institutional upper limit of normal
* Alanine aminotransferase (ALT) =< 2x institutional upper limit of normal
* Aspartate aminotransferase (AST) =< 2x institutional upper limit of normal
* Human immunodeficiency virus (HIV)-1/HIV-2 negative
* Hepatitis B and hepatitis C negative
* The effects of RG1-VLP vaccination on the developing human fetus at the proposed doses are unknown. For this reason, all women of childbearing potential will have a pregnancy test and all heterosexually active women must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* The following persons are not considered to be able to bear children and are therefore eligible to participate without the use of concurrent birth control:

  * Female with bilateral oophorectomy and/or hysterectomy
  * Female with fallopian tubes cut, tied or sealed
  * Female with sterilization implant (e.g. Adiana, Essure) placed > 3 months prior to randomization
  * Female post-menopausal (> 1 year since last menses or prior laboratory follicle stimulating hormone [FSH] value per institutional range indicating post-menopausal)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of any of the following:

  * Prior or current genital warts
  * Treatment for anogenital intraepithelial neoplasia (cervical intraepithelial neoplasia [CIN], anal intraepithelial neoplasia [AIN], vaginal intraepithelial neoplasia [VAIN], vulvar intraepithelial neoplasia [VIN])
  * Systemic cancer treatment within the prior year
* History of anaphylaxis to vaccines
* Any prior vaccination with Gardasil, Gardasil-9, or Cervarix or other HPV vaccine
* Receipt of blood products within 3 months of enrollment, or continuing plasma donation
* Participants receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the adjuvant or to RG1-VLP
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements or preclude protocol vaccination
* Pregnant women or actively lactating women are excluded from this study because RG1-VLP is a vaccine with the potential for teratogenic or abortifacient effects
* Planned receipt of any inactivated vaccine in the 2 weeks preceding and the 2 weeks following any trial vaccination
* Planned receipt of any live attenuated vaccine in the 4 weeks preceding and the 4 weeks following any trial vaccination
* Women with a history of bleeding disorders or use of anticoagulants (aspirin is acceptable)
* Had prior medical diagnoses:

  * Rheumatoid arthritis or other auto-immune disease
  * Congenital or acquired immunodeficiency
  * Collagen vascular disease
* Following medical treatments:

  * Current use of immunosuppressive drugs including corticosteroid use (inhaled or topical steroids are permitted)
* Unrecovered major infections and/or surgical procedures

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months post-3rd RG1-virus-like particle (VLP) vaccination/saline injection
  Safety of the three escalating doses of RG1-VLP will be assessed by adverse events in terms of severity grade and attribution to vaccination as ordinal outcomes. All toxicities will be tabulated and frequencies and percentages of events will be presented for each vaccine dose cohort. The severity of the adverse events will be assessed using the Common Terminology Criteria for Adverse Events 5.0 and supplemented by Food and Drug Administration "Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials."

SECONDARY OUTCOMES:
Determination of serum antibody responses to both human papillomavirus (HPV)16 L1 VLP and to HPV16 L2 | At months 0, 1, 2, 3, 6, 7, and 12
  Will be tested for IgG against HPV16 L1 using a VLP-based enzyme-linked immunosorbent assay (ELISA). The HPV16 L2 17-36 peptide will be synthesized and used for an L2 ELISA. A dose response relationship for log antibody response will be tested with a linear mixed model. Will be summarized with frequency and relative frequencies along with 95% confidence intervals by time, vaccine dose group, and visit. As appropriate, Jonckheere-Terpstra or Cochran-Armitage tests will be used to test for dose-response relationships.
Determination of whether vaccination-induced serum antibody response neutralizes HPV16 | At months 0, 1, 2, 3, 6, 7, and 12
  In vitro HPV pseudovirion (PsV) neutralization assays will be performed for HPV16 and HPV18 and additional PsV types requested by the National Cancer Institute, using an assay specifically developed for sensitivity to L2-specific as well as L1-specific neutralizing antibodies. A dose response relationship with serum neutralizing antibody titer will be tested with linear mixed models or Jonckheere-Terpstra tests as appropriate. Will be summarized with frequency and relative frequencies along with 95% confidence intervals by time, vaccine dose group, and visit. As appropriate, Cochran-Armitage tests will be used to test for dose-response relationships.

OTHER OUTCOMES:
Determination of whether vaccination-induced serum antibody response broadly neutralizes high-risk (hr)HPV other than HPV16 | At months 0, 1, 2, 3, 6, 7 and 12
  A dose response relationship with serum neutralizing antibody titer will be tested with linear mixed models or Jonckheere-Terpstra tests as appropriate.
Determination of whether vaccination induces a cell-mediated immune response | At months 0, 1, and 7
  Peripheral blood mononuclear cells will be isolated. There will be five mice for each human subject. The presence or absence of a vaccination serum antibody response will be recorded for each mouse. A dose-response relationship for serum antibody response will be tested with a repeated measures logistic regression analysis, accounting for the repetition of mice per subject.
Determination of whether vaccination-induced serum antibody response upon passive transfer to naive animals, protects mice against hrHPV pseudovirion challenge | At months 0 and 7
  There will be five mice for each human subject. The presence or absence of a vaccination serum antibody response will be recorded for each mouse. A dose-response relationship for serum antibody response will be tested with a repeated measures logistic regression analysis, accounting for the repetition of mice per subject.
Determination of whether vaccination results in changes in antibody titers in vaginal and oral secretions (via oral rinse), and the effects of vaccination on HPV types in optionally-collected vaginal and oral secretions and eyebrow hair samples | Between months 0, 7 and 12
  These samples will be submitted for future research related to investigating local antibody responses and HPV deoxyribonucleic acid detection.
Safety of administration of Gardasil-9 in individuals post-administration of RG1-VLP | Up to 14 days post-3rd Gardasil-9 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Kirnbauer, Principal Investigator — Medical University of Vienna
Locations (5):
- United States (4):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Staten Island University Hospital, Staten Island, New York
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm